CLINICAL TRIAL: NCT02380742
Title: Topical Anesthetic Use In Pessary Management: A Randomized Double Blinded Placebo Controlled Trial
Brief Title: Topical Anesthetic Use In Pessary Management
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Cynthia Brincat, Assistant Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 206945
Record Dates: First submitted 2015-02-26; First posted 2015-03-05 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Pain
Keywords: Pessary; Pain; EMLA; lidocaine; prilocaine
MeSH Terms: conditions — Pain | interventions — Lidocaine, Prilocaine Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- lidocaine-prilocaine (Experimental): 4 mL of lidocaine-prilocaine cream
  Interventions: Drug: lidocaine-prilocaine cream
- Placebo (Placebo Comparator): 4 mL of placebo cream
  Interventions: Drug: Placebo cream

INTERVENTIONS:
Drug: lidocaine-prilocaine cream — The patient will then be positioned in dorsal lithotomy position with the use of stirrups. Two mL of EMLA cream will be placed into the vagina and 2 mL will be spread on the perineum. The cream placed into the vagina will be introduced to the level of the pessary with the practitioners' finger. Once application is completed, a timer will be set for five minutes. After five minutes, the patient will again be placed into dorsal lithotomy position with the use of stirrups. The pessary will be removed per practitioners' usual practice. The patient will be asked to mark her pain score for at this point
  Other Names: 5% EMLA cream
  Arms: lidocaine-prilocaine
Drug: Placebo cream — The patient will then be positioned in dorsal lithotomy position with the use of stirrups. Two mL of placebo cream will be placed into the vagina and 2 mL will be spread on the perineum. The cream placed into the vagina will be introduced to the level of the pessary with the practitioners' finger. Once application is completed, a timer will be set for five minutes. After five minutes, the patient will again be placed into dorsal lithotomy position with the use of stirrups. The pessary will be removed per practitioners' usual practice. The patient will be asked to mark her pain score for at this point
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate if lidocaine-prilocaine (EMLA 5%) cream can reduce pain and discomfort at the time of vaginal pessary removal and insertion. Half of the participants will receive lidocaine-prilocaine (EMLA 5%) cream and the other half will receive a placebo cream.

DETAILED DESCRIPTION:
Lidocaine-prilocaine (EMLA 5%) cream has been shown to be effective in reducing pain during minor gynecologic procedures. The primary objective of this trial is to determine if the use of 5% EMLA cream at the time of pessary removal and insertion reduces pain when compared to the use of placebo cream.

Participants will be randomized to receive either 10 grams of 5% EMLA cream (4 mL) or 4 mL of placebo cream (aqueous cream BP). Cream will be applied in office at the time of pessary removal and insertion.

ELIGIBILITY:
Inclusion Criteria:

* Women in the Loyola Urogynecology clinic who use a pessary for management of pelvic organ prolapse (POP) or urinary incontinence (UI)
* Read and speak the English language

Exclusion Criteria:

* Non-English speaking
* Allergy or contraindication to topical anesthetic
* Participation/randomization in the study at a previous visit
* Currently pregnant or lactating or planning a pregnancy within the next 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Brincat, MD, Principal Investigator — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Nygaard I, Bradley C, Brandt D; Women's Health Initiative. Pelvic organ prolapse in older women: prevalence and risk factors. Obstet Gynecol. 2004 Sep;104(3):489-97. doi: 10.1097/01.AOG.0000136100.10818.d8. PMID 15339758
- [Background] Melville JL, Katon W, Delaney K, Newton K. Urinary incontinence in US women: a population-based study. Arch Intern Med. 2005 Mar 14;165(5):537-42. doi: 10.1001/archinte.165.5.537. PMID 15767530
- [Background] Olsen AL, Smith VJ, Bergstrom JO, Colling JC, Clark AL. Epidemiology of surgically managed pelvic organ prolapse and urinary incontinence. Obstet Gynecol. 1997 Apr;89(4):501-6. doi: 10.1016/S0029-7844(97)00058-6. PMID 9083302
- [Background] Donnelly MJ, Powell-Morgan S, Olsen AL, Nygaard IE. Vaginal pessaries for the management of stress and mixed urinary incontinence. Int Urogynecol J Pelvic Floor Dysfunct. 2004 Sep-Oct;15(5):302-7. doi: 10.1007/s00192-004-1163-7. Epub 2004 Aug 5. PMID 15300365
- [Background] Nguyen JN, Jones CR. Pessary treatment of pelvic relaxation: factors affecting successful fitting and continued use. J Wound Ostomy Continence Nurs. 2005 Jul-Aug;32(4):255-61; quiz 262-3. doi: 10.1097/00152192-200507000-00010. PMID 16030465
- [Background] Lone F, Thakar R, Sultan AH, Karamalis G. A 5-year prospective study of vaginal pessary use for pelvic organ prolapse. Int J Gynaecol Obstet. 2011 Jul;114(1):56-9. doi: 10.1016/j.ijgo.2011.02.006. Epub 2011 May 14. PMID 21575953
- [Background] Keskin AE, Onaran Y, Duvan IC, Simavli S, Kafali H. Topical anesthetic (lidocaine-prilocaine) cream application before speculum examination in postmenopausal women. J Minim Invasive Gynecol. 2012 May-Jun;19(3):350-5. doi: 10.1016/j.jmig.2012.01.005. Epub 2012 Mar 13. PMID 22417905
- [Background] Zilbert A. Topical anesthesia for minor gynecological procedures: a review. Obstet Gynecol Surv. 2002 Mar;57(3):171-8. doi: 10.1097/00006254-200203000-00022. PMID 11889416
- [Background] Wahlgren CF, Lillieborg S. Split-skin grafting with lidocaine-prilocaine cream: A meta-analysis of efficacy and safety in geriatric versus nongeriatric patients. Plast Reconstr Surg. 2001 Mar;107(3):750-6. doi: 10.1097/00006534-200103000-00015. PMID 11304601
- [Derived] Taege SK, Adams W, Mueller ER, Brubaker L, Fitzgerald CM, Brincat C. Anesthetic Cream Use During Office Pessary Removal and Replacement: A Randomized Controlled Trial. Obstet Gynecol. 2017 Jul;130(1):190-197. doi: 10.1097/AOG.0000000000002098. PMID 28594757

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lidocaine-prilocaine | Placebo
Started | 28 | 26
Completed | 27 | 26
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidocaine-prilocaine | Placebo | Total
Number analyzed (Participants) | 27 | 26 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.64 (10.43) | 79.95 (8.01) | 77.76 (9.49)
Gender [Count of Participants; unit: Participants]
  Female | 27 | 26 | 53
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 23 | 24 | 47
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 25 | 22 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5
BMI, Continuous [Mean (Standard Deviation); unit: kg/m^2] | 28.11 (6.06) | 29.47 (6.59) | 28.78 (6.30)
Median gravidity (IQR) [Median (Inter-Quartile Range); unit: number of pregnancies] | 3 [2 to 4] | 3 [2 to 4] | 3 [2 to 4]
Median parity (range) [Median (Inter-Quartile Range); unit: number of viable pregnancies] | 3 [2 to 4] | 3 [2 to 4] | 3 [2 to 4]
Median pessary months (IQR) [Median (Inter-Quartile Range); unit: months] | 18 [6 to 26] | 14 [5 to 32] | 15 [6 to 26]
Median pessary size (IQR) [Median (Inter-Quartile Range); unit: mm] | 70 [64 to 76] | 70 [65 to 76] | 70 [64 to 76]
Reason for pessary [Number; unit: participants]
  Prolapse | 14 | 15 | 29
  Incontinence | 7 | 1 | 8
  Prolapse & Incontinence | 6 | 10 | 16
Type of pessary [Number; unit: participants]
  Gelhorn | 0 | 5 | 5
  Ring | 3 | 1 | 4
  Ring with support | 13 | 10 | 23
  Incontinence ring | 2 | 1 | 3
  Incontinence dish | 4 | 4 | 8
  Incontinence dish with support | 5 | 5 | 10
Vaginal erosions [Number; unit: participants]
  No | 25 | 23 | 48
  Yes | 2 | 3 | 5
Weekly topical estrogen [Number; unit: participants]
  No | 20 | 16 | 36
  Yes | 7 | 10 | 17
Menopausal status [Number; unit: participants]
  Premenopausal | 0 | 0 | 0
  Postmenopausal | 27 | 26 | 53
Mean age at menopause (SD) [Mean (Standard Deviation); unit: years] | 48.67 (5.92) | 49.10 (6.85) | 48.88 (6.33)
Prior hysterectomy [Number; unit: participants]
  No | 16 | 19 | 35
  Yes | 11 | 7 | 18
Sexually active [Number; unit: participants]
  No | 23 | 26 | 49
  Yes | 4 | 0 | 4
Pain with intercourse [Number; unit: participants]
  No | 12 | 9 | 21
  Yes | 0 | 0 | 0
  Not applicable | 15 | 17 | 32
Tobacco use [Number; unit: participants]
  No | 26 | 24 | 50
  Yes | 1 | 2 | 3
Pessary satisfaction [Number; unit: participants]
  Dissatisfied | 0 | 0 | 0
  Somewhat dissatisfied | 0 | 1 | 1
  Neutral | 1 | 0 | 1
  Somewhat satisfied | 4 | 6 | 10
  Very satisfied | 22 | 19 | 41
Baseline VAS scores [Mean (Standard Deviation); unit: units on a scale] — The Visual Analogue Scale (VAS) consists of a 10-cm-long straight line, scaled from 0 to 10 (0 = no pain and 10 = severe pain) without numerical values on the scale, except for 0 and 10.
  units on a scale
    Mean paper form | 0.29 (0.73) | 0.23 (0.48) | 0.26 (0.61)
    Mean electronic form | 0.51 (0.69) | 0.52 (0.51) | 0.52 (0.60)

OUTCOME MEASURES:

1. Primary Outcome: VAS Score at the Time of Pessary Removal Adjusting for Baseline Pain
Description: Self-reported pain intensity at time of pessary removal controlling for baseline pain. Scale is from 0 to 10 (0=no pain and 10=worst pain)
Time Frame: Removal of Pessary
Measure: Least Squares Mean (Standard Error); unit: Centimeters
Arm/Group | Lidocaine-prilocaine | Placebo
Number analyzed (Participants) | 27 | 26
Centimeters | 1.76 (0.57) | 3.81 (0.58)
Statistical Analysis 1: Comparison: Lidocaine-prilocaine vs Placebo; The null hypothesis was that patients' pain scores at removal were the same between the lidocaine and placebo groups after controlling for baseline pain; Test type: Superiority or Other; p = .02, ANCOVA; Mean Difference (Final Values) = 2.87, Standard Error of Mean 0.47

2. Secondary Outcome: VAS Score at the Time of Pessary Removal Adjusting for Pessary Type and Investigator Training
Description: Self-reported pain intensity at time of pessary removal after controlling for pessary type and investigator training level. Scale is from 0 to 10 centimeters (0=no pain and 10=worst pain)
Time Frame: Removal of Pessary
Measure: Least Squares Mean (Standard Error); unit: Centimeters
Arm/Group | Lidocaine-prilocaine | Placebo
Number analyzed (Participants) | 27 | 26
Centimeters | 1.81 (0.59) | 3.76 (0.60)
Statistical Analysis 1: Comparison: Lidocaine-prilocaine vs Placebo; The null hypothesis was that patients' pain scores at removal were the same between the lidocaine and placebo groups after controlling for investigator training and pessary type; Test type: Superiority or Other; p = .03, ANCOVA; Mean Difference (Final Values) = -1.96, Standard Error of Mean 0.87

3. Secondary Outcome: VAS Score at the Time of Pessary Removal Adjusting for Baseline Pain and Patient Age
Description: Self-reported pain intensity at time of pessary removal after controlling for patient age and baseline pain score. Scale is from 0 to 10 centimeters (0=no pain and 10=worst pain)
Time Frame: Removal of Pessary
Measure: Least Squares Mean (Standard Error); unit: Centimeters
Arm/Group | Lidocaine-prilocaine | Placebo
Number analyzed (Participants) | 27 | 26
Centimeters | 1.88 (0.58) | 3.69 (0.59)
Statistical Analysis 1: Comparison: Lidocaine-prilocaine vs Placebo; The null hypothesis was that patients' pain scores at removal were the same between the lidocaine and placebo groups after controlling for baseline pain and patient age; Test type: Superiority or Other; p = .03, ANCOVA; Mean Difference (Final Values) = -1.811, Standard Error of Mean 0.83

4. Secondary Outcome: VAS Score at the Time of Pessary Insertion Adjusting for Baseline Pain
Description: Practitioner's perception of patient's pain score at time of pessary insertion adjusting for baseline pain. Scale is from 0 to 10 centimeters (0=no pain and 10=worst pain)
Time Frame: Insertion of Pessary
Population: After baseline and removal study activities were recorded, one of the patients in the placebo group was withdrawn by the investigator due to vaginal erosion.
Measure: Least Squares Mean (Standard Error); unit: Centimeters
Arm/Group | Lidocaine-prilocaine | Placebo
Number analyzed (Participants) | 27 | 25
Centimeters | 0.61 (0.43) | 1.68 (0.44)
Statistical Analysis 1: Comparison: Lidocaine-prilocaine vs Placebo; The null hypothesis was that patients' pain scores at insertion were the same between the lidocaine and placebo groups after controlling for baseline pain; Test type: Superiority or Other; p = .09, ANCOVA; Mean Difference (Final Values) = -1.07, Standard Error of Mean 0.63

ADVERSE EVENTS:
Time Frame: Reported adverse events includes events from initial enrollment to study completion.
Arm/Group | Lidocaine-prilocaine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/26
Other Adverse Events (participants affected / at risk) | 0/27 | 0/26

LIMITATIONS AND CAVEATS:
There are no limitations or caveats to report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes